CLINICAL TRIAL: NCT03564015
Title: Smartphone App to Improve Functional Outcomes in Children With Acute Ankle Inversion Injuries: a Randomized Controlled Trial
Brief Title: Smartphone App to Improve Functional Outcomes in Ankle Sprains
Acronym: SPRAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The intervention (guidance recovery app) was malfunctioning and not storing data for efficacy outcomes.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111817
Record Dates: First submitted 2018-04-09; First posted 2018-06-20 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized, open-label, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone app (Experimental): The smartphone group will not be given paper-based discharge instructions in the ED. They will download onto their smartphone device an Intervention App that will allow recording of the above mentioned study outcomes and contains an interactive educational component encompassing the identical information outlined in the paper handout. The app will provide educational guidance towards recovery using a feedback algorithm that will recommend on a daily basis, the use of ice, elevation, range of motion exercises, and/or analgesics based on the participant's report of their pain using the FPS-R.
  Interventions: Other: Smartphone app
- Paper handout (Active Comparator): The paper handout group will be asked to read the paper-based discharge instructions in the ED, outlining pharmacological and non-pharmacological pain management and return to activity. They will download onto their smartphone device a Recording App that will only allow them to record the following study outcome measures: daily use of ice, analgesia, range of motion exercises, elevation, pain using the Faces Pain Scale - Revised (FPS-R), and ASKp scores on days 3, 5, 7, 10, 12, and 14.
  Interventions: Other: Paper handout

INTERVENTIONS:
Other: Smartphone app — Apple or Android app to provide education to guide functional recovery and allow recording of pain, management, and functional outcome using the Activities Scale for Kids performance version (ASKp) at home
  Arms: Smartphone app
Other: Paper handout — Paper handout to guide functional recovery. Also includes a version of the smartphone app described above that only allows recording of pain, functional outcome, and management at home.
  Arms: Paper handout

SUMMARY:
Ankle sprains are the most common musculoskeletal complaint of children presenting to the emergency department (ED). Healing can often be protracted, leading to prolonged pain, missed school and work, and delayed return to a normal activity level. Smartphone apps have been shown to be associated with greater caregiver knowledge and improved outcomes in a number of conditions but have not been explored in ankle sprains. The investigators would like to know if using a smartphone app for children with ankle inversion injuries leads to improved functional outcomes such as pain, mobility, and return to activity. The investigators will be comparing a smartphone app that provides education and daily management reminders to a paper handout to see if the former leads to improved functional recovery.

DETAILED DESCRIPTION:
Comprehensive discharge instructions are an integral part of care children discharged from the emergency department (ED). Unfortunately, providing consistent and thorough discharge instructions is highly limited by the workflow constraints of a busy ED. Currently, paper instructions are the standard for providing ED discharge information. Yet, there remains a great deal of variety in delivery of discharge instructions (1) and there is evidence that patients often do not fully comprehend (2, 3), recall (4), nor comply (5) with discharge instructions. Consequently, caregivers often commit errors related to knowledge and execution of ED discharge instructions (6). The use of a smartphone app following discharge from the ED offers a potential means to improve adherence to discharge instructions through consistent information, simplification of content, and reminders (2). Acute ankle sprains are one of the most common complaints presenting to primary care offices and EDs (7). In Canada and the United States, there are more than 2 million ED visits annually due to ankle trauma in children; 85% due to forced inversion (8). Adolescents and young adults have the highest incidence of ankle sprain (7.2 per 1,000 person-years). Although ankle sprains are often perceived as minor injuries, they can have a highly variable prognosis, with up to 64% of patients failing to achieve full recovery (9). Current guidelines are limited in determining prognostic factors associated with functional recovery (9). The resulting 'one-size fits all' approach (controlling acute inflammatory symptoms (9), using cryotherapy and anti-inflammatory medications, and early mobilization (7)) fails to consider the grade of injury, baseline level of functioning, and individual pain tolerance of the child. Educational guidance individualized to pain beyond the ED may improve functional outcomes. As of 2015, 82% of people age 18-49 years owned an app-enabled smartphone, and over half (58%) download health related smartphone apps (10). In adult medicine, many health-related smartphone apps have been shown to be associated with greater caregiver knowledge and improved outcomes in allergic rhinitis (10), post-operative monitoring (11), and musculoskeletal conditions (12). In children and adolescents, several studies have explored smartphone apps for asthma (13) and diabetes (14, 15). To date however, no smartphone apps have been developed for acute musculoskeletal injury management in children.

ELIGIBILITY:
Inclusion Criteria:

(i) Age 12-21 years (ii) Presenting to the Emergency Department of the Children's Hospital, London Health Sciences Centre, London, Ontario, with a unilateral acute (<48 hours) ankle inversion injury.

(iii) Use a WiFi enabled smartphone with either an iOS or Android operating system with enough memory capability to host the App.

The diagnosis of an ankle inversion injury will be made on a clinical basis by the treating emergency physician after a fracture has been ruled out radiographically. We will include all grades of ankle injuries, including suspected Salter-Harris I of the distal tibia or fibula.

Exclusion Criteria:

* Children unable to read or understand English above at least a grade 8 literacy level
* Children who are not independently ambulatory (without the use of an assistive device)
* Children with a developmental disability precluding the full comprehension of study-related procedures,
* Children with multi-system or multi-limb injuries
* Children with a concomitant lower extremity fracture or dislocation (with the exception of a suspected Salter-Harris type I injury).

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Activities Scale for Kids performance version (ASKp) | Day 14 +/- 1 day post-discharge
  30 item self-report questionnaire on functional performance with total score ranging from 0-100 with higher values representing greater function

SECONDARY OUTCOMES:
Activities Scale for Kids performance version (ASKp) | Day 3, 5, 7, 10, and 12 +/- 1 day post-discharge
  30 item self-report questionnaire on functional performance with total score ranging from 0-100 with higher values representing greater function
Time to return to baseline ASKp score | Days 1-14 post discharge
  30 item self-report questionnaire on functional performance with total score ranging from 0-100 with higher values representing greater function
Pain using the Faces Pain Scale - Revised (FPS-R) | Days 1-14 post discharge
  Self-report 6-item ordinal scale ranging from 0-5 with higher score indicating more pain
Use of non-pharmacological measures (ice, compression, other) | Days 1-14 post discharge
  Frequency
Use of pharmacological analgesia (NSAIDs, acetaminophen) | Days 1-14 post discharge
  Frequency

CONTACTS AND LOCATIONS:
Overall Officials: Janet Knechtel, BA, Study Chair — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No